CLINICAL TRIAL: NCT00447031
Title: Intravitreal Bevacizumab Combined With Intravitreal Triamcinolone Acetonide Injection Versus Intravitreal Bevacizumab for Age Related Macular Degeneration
Brief Title: Combination Therapy for Neovascular Age Related Macular Degeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patients who met inclusion criteria
Sponsor: Yonsei University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: koh02
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2009-03

CONDITIONS: Macular Degeneration
Keywords: age related macular degeneration; intravitreal bevacizumab; intravitreal triamcinolone acetonide; neovascular age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intravitreal bevacizumab and triamcinolone acetonide

SUMMARY:
Exudative age related macular degeneration (ARMD) is most common cause of blindness in old population. It is clear that no single therapy addresses the multifactorial pathogenesis of the disease. Recently, studies of intravitreal anti-VEGF therapies such as pegaptanib and bevacizumab have shown the beneficial effect in visual acuity in the treatment of neovascular ARMD. However, the problem with these intravitreal injections is that therapy must be frequently administered for a prolonged but unknown period of time to maintain the benefit. Prolonged, frequent injections may be associated with additional safety risk,lack of convenience and high treatment cost.

Intravitreal steroid injection with anti-inflammatory properties limits any further VEGF upregulation initiated by the inflammation which has been known as one of the pathogenesis and causes of recurrence after the treatment of the neovascular ARMD.

The researchers hypothesize that the combined treatment of intravitreal bevacizumab and triamcinolone acetonide may decrease the recurrence rate after the treatment and obviate the frequent intravitreal injections in the treatment of neovascular ARMD.

In this study, the researchers will compare the recurrence rate of combined treatment of intravitreal bevacizumab and triamcinolone acetonide versus intravitreal bevacizumab alone in the treatment of neovascular ARMD.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular ARMD confirmed with 90+ noncontact lens biomicroscopy, fluorescein angiography, ocular coherence tomography

Exclusion Criteria:

* Intractable systemic hypertension
* Recent myocardial infarct within 6 months at enrollment
* Recent cerebrovascular attack within 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
recurrence rate
best corrected visual acuity

SECONDARY OUTCOMES:
complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jun Koh, Principal Investigator — YUMC
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Costa RA, Jorge R, Calucci D, Melo LA Jr, Cardillo JA, Scott IU. Intravitreal bevacizumab (Avastin) in combination with verteporfin photodynamic therapy for choroidal neovascularization associated with age-related macular degeneration (IBeVe Study). Graefes Arch Clin Exp Ophthalmol. 2007 Sep;245(9):1273-80. doi: 10.1007/s00417-007-0557-x. Epub 2007 Feb 28. PMID 17333238
- [Background] Augustin AJ, Puls S, Offermann I. Triple therapy for choroidal neovascularization due to age-related macular degeneration: verteporfin PDT, bevacizumab, and dexamethasone. Retina. 2007 Feb;27(2):133-40. doi: 10.1097/IAE.0b013e3180323de7. PMID 17290193
- [Background] Dhalla MS, Shah GK, Blinder KJ, Ryan EH Jr, Mittra RA, Tewari A. Combined photodynamic therapy with verteporfin and intravitreal bevacizumab for choroidal neovascularization in age-related macular degeneration. Retina. 2006 Nov-Dec;26(9):988-93. doi: 10.1097/01.iae.0000247164.70376.91. PMID 17151484
- [Background] Aisenbrey S, Ziemssen F, Volker M, Gelisken F, Szurman P, Jaissle G, Grisanti S, Bartz-Schmidt KU. Intravitreal bevacizumab (Avastin) for occult choroidal neovascularization in age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2007 Jul;245(7):941-8. doi: 10.1007/s00417-006-0471-7. Epub 2006 Dec 21. PMID 17186262
- [Background] Gomi F, Nishida K, Oshima Y, Sakaguchi H, Sawa M, Tsujikawa M, Tano Y. Intravitreal bevacizumab for idiopathic choroidal neovascularization after previous injection with posterior subtenon triamcinolone. Am J Ophthalmol. 2007 Mar;143(3):507-10. doi: 10.1016/j.ajo.2006.10.050. Epub 2006 Dec 8. PMID 17317397
- [Background] Jonas JB, Libondi T, Ihloff AK, Harder B, Kreissig I, Schlichtenbrede F, Sauder G, Spandau UH. Visual acuity change after intravitreal bevacizumab for exudative age-related macular degeneration in relation to subfoveal membrane type. Acta Ophthalmol Scand. 2007 Aug;85(5):563-5. doi: 10.1111/j.1600-0420.2007.00891.x. Epub 2007 Feb 27. PMID 17324219